CLINICAL TRIAL: NCT06161428
Title: Optical Guided Sentinel Node Biopsy for Staging of Vulvar Cancer ( SENTIVUC II)
Brief Title: Optical Guided Sentinel Node Biopsy for Staging of Vulvar Cancer
Acronym: SENTIVUC II
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Ligita Paskeviciute Froding, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: P-2022-946
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Vulva Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the feasibility of applying the SLN mapping technique in combination with FDG-PET/CT imaging in women with vulva cancer tumour size >4 cm, multifocal tumors and local recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vulva cancer, tumor > 4 cm, multifocal tumor, or local recurrences in vulva

Exclusion Criteria:

* Previous external irradiation of the vulva or groins
* Former sentinel node or inguinal lymphadenectomy in the relevant groin
* Known allergy to ICG or iodine
* Patient is in active treatment for other cancer and/or disseminated disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or recurrent vulva cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Three years
  Sensitivity of sentinel lymph node mapping

SECONDARY OUTCOMES:
Negative predictive value | Three years
  Negative predictive value of sentinel lymph node mapping

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Copenhagen, Denmark